CLINICAL TRIAL: NCT05673343
Title: The Prognostic Impact Of The Neutrophil To Lymphocyte Ratio In Patients With Locally Advanced Rectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shymaa tarek shafea, The Prognostic Impact Of The Neutrophil To Lymphocyte Ratio In Patients with Locally Advanced Rectal Cancer, Assiut University
Other Study IDs: Locally advanced rectal cancer
Record Dates: First submitted 2023-01-04; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: the Prognostic Value of Pre-treatment NLR in Patients With Locally Advenced Rectal Cancer and Post-treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Complete blood count: Complete blood count with differential should be done within 2 weeks before starting CCRT. We will calculate NLR as total neutrophilic count divided by total lymphocytic count for each patient before starting the treatment.
  Two protocols of the treatment: first is by starting with CCRT then surgery (Total Neoadjuvant Therapy), second is CCRT then surgery then continue chemotherapy: FOLFOX , Xeloda or CAPOX.
  Radiotherapy dose: long course radiation therapy at the dose of 45 to 50 Gray (Gy) in 25 to 28 fractions to the pelvis by NCCN recommendation. Short-course radiation therapy (25 Gy in 5 fractions).
  Patients should be kept on follow up after complete their treatment every three months till disease progression occur, death of the patient or at least 12 months of follow up.

SUMMARY:
In this study, we aim to investigate the prognostic value of pre-treatment NLR in patients with locally advenced rectal cancer and post-treatment

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common malignancy and the second leading cause of cancer-related death worldwide.[1] Rectal cancer accounts for 30% to 35% of CRCs[2], Between 5% and 10% of patients with rectal cancer present with locally advanced rectal cancer (LARC),[3] Useful and practical prognostic biomarkers obtained before treatment are anticipated to predict the outcome after main treatment. Such biomarkers will help in planning strategies for adjustment of postoperative adjuvant therapy.[4]

Inflammation-induced markers play an important role in tumorigenesis and tumor progression. More evidences had reported systemic inflammation-based biomarkers could be used to predict tumor behavior.[4] Two convenient and economic measures of systemic inflammation, neutrophil-to-lymphocyte ratio (NLR) and platelet-to-lymphocyte ratio (PLR), that reflect the interaction between inflammation and host immune status, making them potential prognostic factors for various types of cancers. Increased NLR has been advocated to be an independent prognostic factor for poor survival outcomes in pancreatic cancer, CRC, and gastric cancer [5-6].

In this study, we aim to investigate the prognostic value of pre-treatment NLR in patients with locally advenced rectal cancer and post-treatment

ELIGIBILITY:
Inclusion Criteria:

- Patients aged 18-year-old or more 2-Histopathologically proved to be rectal carcinoma. 3- locally advanced stage II and stage III according to AJCC TNM staging 8th edition 4- fit for concurrent chemoradiation therapy (CCRT) with adequate organ function.

5- Performance status 0-1 according to ECOG PS

Exclusion Criteria:

* 1- metastatic disease 2- Younger than 18 year old 3-Any other malignancy 4-There is contraindication for CCRT

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-year-old or more 2-Histopathologically proved to be rectal carcinoma. 3- locally advanced stage II and stage III according to AJCC TNM staging 8th edition 4- fit for concurrent chemoradiation therapy (CCRT) with adequate organ function.
  5- Performance status 0-1 according to ECOG PS
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-04 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
disease free-survival | 2-5 yrs
  defined as the time from the day of disease diagnosis until the day of disease failure.

SECONDARY OUTCOMES:
overall survival (OS | 2-5 years
  defined as the time from the day of disease diagnosis until the date of death.

REFERENCES:
- [Background] Yang G, Chang JS, Choi JE, Baek ES, Kim SS, Byun HK, Cho Y, Koom WS, Yang SY, Min BS, Shin SJ. Association of neutrophil-to-lymphocyte ratio, radiotherapy fractionation/technique, and risk of development of distant metastasis among patients with locally advanced rectal cancer. Radiat Oncol. 2022 May 21;17(1):100. doi: 10.1186/s13014-022-02065-8. PMID 35597954
- [Background] Nagasaki T, Akiyoshi T, Fujimoto Y, Konishi T, Nagayama S, Fukunaga Y, Ueno M. Prognostic Impact of Neutrophil-to-Lymphocyte Ratio in Patients with Advanced Low Rectal Cancer Treated with Preoperative Chemoradiotherapy. Dig Surg. 2015;32(6):496-503. doi: 10.1159/000441396. Epub 2015 Nov 7. PMID 26544755
- [Background] Sun Y, Zhang Y, Huang Z, Lin H, Lu X, Huang Y, Chi P. Combination of Preoperative Plasma Fibrinogen and Neutrophil-to-Lymphocyte Ratio (the F-NLR Score) as a Prognostic Marker of Locally Advanced Rectal Cancer Following Preoperative Chemoradiotherapy. World J Surg. 2020 Jun;44(6):1975-1984. doi: 10.1007/s00268-020-05407-3. PMID 32020327
- [Background] Cha YJ, Park EJ, Baik SH, Lee KY, Kang J. Prognostic impact of persistent lower neutrophil-to-lymphocyte ratio during preoperative chemoradiotherapy in locally advanced rectal cancer patients: A propensity score matching analysis. PLoS One. 2019 Mar 22;14(3):e0214415. doi: 10.1371/journal.pone.0214415. eCollection 2019. PMID 30901357
- [Result] Toiyama Y, Inoue Y, Kawamura M, Kawamoto A, Okugawa Y, Hiro J, Saigusa S, Tanaka K, Mohri Y, Kusunoki M. Elevated platelet count as predictor of recurrence in rectal cancer patients undergoing preoperative chemoradiotherapy followed by surgery. Int Surg. 2015 Feb;100(2):199-207. doi: 10.9738/INTSURG-D-13-00178.1. PMID 25692418